CLINICAL TRIAL: NCT04173611
Title: Phase 1, Randomized, Double-Blind, Active and Placebo Controlled, Dose Escalation Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of EXPAREL® Administered Via a Single Intrathecal Injection to Healthy Volunteers.
Brief Title: Evaluation of Safety, Pharmacokinetics and Pharmacodynamics of EXPAREL® Administered Via a Single Intrathecal Injection to Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated for strategic and administrative reasons
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 402-C-121
Record Dates: First submitted 2019-11-18; First posted 2019-11-22 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: Pharmacodynamics; Pharmacokinetics; Safety; Efficacy
MeSH Terms: interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The decision to proceed to each next cohort will be made following a full review of the safety, PK, and PD data from the previous completed cohort(s).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each of the cohorts will be masked as to proceed to subsequent next dose escalation cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EXPAREL® (Experimental): For those subjects randomized to EXPAREL® arm - the dose of EXPAREL® will be determined by the cohort. Starting at 1mL (13.3mg) for cohort 1, the volume of EXPAREL® will be increased by 1 mL in each subsequent cohort for a maximum of 4mL (53.2mg).
  Interventions: Drug: EXPAREL
- Bupivacaine (Active Comparator): In each cohort, subjects randomized to the bupivacaine arm will receive 15mg of plain bupivacaine HCL (the equivalent of 13.3mg bupivacaine base) providing a 1:1 reference to the starting dose level chosen for EXPAREL®.
  Interventions: Drug: Bupivacaine Hydrochloride
- Placebo (Active Comparator): Subjects in the placebo arm will receive normal saline intrathecal injection
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: EXPAREL — Injection into the Intrathecal space.
  Arms: EXPAREL®
Drug: Bupivacaine Hydrochloride — Injection into the Intrathecal space.
  Other Names: 0.5% Bupivacaine HCl
  Arms: Bupivacaine
Other: Placebo — Injection into the Intrathecal space.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Primary objective: To assess the safety and tolerability of EXPAREL® administered as a single intrathecal injection in healthy volunteers

Secondary objective: To characterize the pharmacokinetic (PK) and pharmacodynamic (PD) profile of EXPAREL® administered as a single intrathecal injection in healthy volunteers

DETAILED DESCRIPTION:
This is a Phase-1, single center, randomized, double-blind, active and placebo-controlled study in approximately 40 healthy adult subjects.

On Day 1, eligible subjects will be randomized in blocks of 5, in a ratio of 3:1:1 to receive EXPAREL® or bupivacaine or placebo (saline) injection, respectively. Starting with treatment Cohort 1, healthy volunteers will be randomized to the 3 treatment arms within cohorts. Each cohort will consist of 10 subjects (6 EXPAREL®, 2 bupivacaine and 2 placebo). In each cohort, all 10 subjects in each cohort will receive cerebrospinal fluid (CSF) taps. Within the EXPAREL® arm, subjects will be randomized 2:1 with 4 subjects undergoing CSF tap and 2 subjects not undergoing CSF tap in each cohort. Subjects who are not undergoing CSF tap, will still be injected with needles without draw of CSF to prevent subject bias. Such a randomization will allow for characterization of the complete pharmacodynamics profile of the drug without risk of drug removal in the CSF. For those subjects randomized to the EXPAREL® arm - the dose of EXPAREL® will be determined by the cohort. Starting at 1 mL (13.3 mg) for Cohort 1, the volume of EXPAREL® will be increased by 1 mL in each subsequent cohort for a maximum of 4 mL (53.2 mg). The decision to proceed to the next cohort will be made following a full review of the safety, PK, and PD (sensory and motor) data from current completed cohort(s). All subjects will remain in the EPRU for 5 days after drug administration and will be discharged on Day 6. Subjects will be instructed to return for a follow up visit on Day 9. Adverse events (AEs) and serious adverse events (SAEs) will be recorded from the time of consent through 30 days after drug administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female volunteers ages ≥18 and ≤50 years old.
2. American Society of Anesthesiologists (ASA) physical status 1.
3. Able to provide informed consent, adhere to the study schedule, and complete all study assessments.

Exclusion Criteria:

1. Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications for which an alternative is not named in the protocol (eg, amide-type local anesthetics, opioids, bupivacaine, non-steroidal anti-inflammatory drugs [NSAIDs], spinal anesthesia).
2. Impaired renal or hepatic function (eg, serum creatinine level >2 mg/dL [176.8 μmol/L], blood urea nitrogen level >50 mg/dL [17.9 mmol/L], serum aspartate aminotransferase [AST] level >1.5 times the upper limit of normal [ULN], or serum alanine aminotransferase [ALT] level >1.5 times the ULN).
3. Subjects at an increased risk for bleeding or who have a coagulation disorder (defined as platelet count less than 80,000 × 103/mm3).
4. Concurrent painful physical condition that may require analgesic treatment (such as long-term, consistent use of opioids) in the post dosing period for pain and which may confound the post dosing assessments.
5. Women of childbearing potential must have a documented negative pregnancy test at screening and must be confirmed on the day of drug administration. If postmenopausal, must have a documented Follicle Stimulating Hormone (FSH) test confirming menopause at screening.
6. Currently pregnant, nursing, or planning to become pregnant during the study or within 30 days after completion of the study.
7. Positive serology test result for Human Immunodeficiency Virus (HIV), Hepatitis B virus, or Hepatitis C virus.
8. Clinically significant abnormal ECG that in the opinion of the investigator would preclude the subject from participation in the study.
9. Previous participation in a Pacira study.
10. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
11. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-versus-time curve | 6-8 weeks
  Pharmacokinetic endpoint
Maximum plasma concentration (Cmax) and time of Cmax (Tmax). | 6-8 weeks
  Pharmacokinetic endpoint
The apparent terminal elimination half-life (t1/2el) | 6-8 weeks
  Pharmacokinetic endpoint
Apparent clearance (CL/F) | 6-8 weeks
  Pharmacokinetic endpoint
Apparent volume of distribution (Vd) | 6-8 weeks
  Pharmacokinetic endpoint

SECONDARY OUTCOMES:
Incidence of treatment-emergent AEs (TEAEs) through Day 9 | 6-8 weeks
  Safety endpoint
Proportion of subjects who have any of neurological events | 6-8 weeks
  Safety endpoint

OTHER OUTCOMES:
Average time to onset of sensory block and motor block | 6-8 weeks
  Pharmacodynamic Endpoint
Average duration of sensory block and motor block | 6-8 weeks
  Pharmacodynamic Endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Donald C Manning, MD, PhD, Study Director — Pacira Pharmaceuticals, Inc
Locations (1):
- Duke University, Durham, North Carolina, United States